CLINICAL TRIAL: NCT01891110
Title: Prevention of Orthostatic Hypotension With Electric Stimulation in Persons With Acute SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-26
Record Dates: First submitted 2013-06-04; First posted 2013-07-02 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Spinal Cord Injury; Orthostatic Hypotension
Keywords: electric stimulation; tilt-table
MeSH Terms: conditions — Spinal Cord Injuries; Hypotension, Orthostatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ES of the abdominal muscles (Experimental): ES with surface electrodes, fixed stimulation parameters and individual mA
  Interventions: Procedure: ES of the abdominal muscles
- ES of limbs & abdomen (Experimental): The combination of the ES of the lower limb muscles and the abdominal muscles.
  Interventions: Procedure: ES of limbs & abdomen
- ES of the limb muscles (Experimental): Lower limb muscles were stimulated to produce a milking mechanism from the distal to proximal part of the limb to pump the venous blood from the peripheral to the central part of the body
  Interventions: Procedure: ES of the limb muscles

INTERVENTIONS:
Procedure: ES of the abdominal muscles — ES was applied with surface electrodes and fixed stimulation parameters with individual mA, depending on each patients´ sensibility.
  Arms: ES of the abdominal muscles
Procedure: ES of the limb muscles — Lower limb muscles were stimulated to produce a milking mechanism from the distal to proximal part of the limb to pump the venous blood from the peripheral to the central part of the body
  Arms: ES of the limb muscles
Procedure: ES of limbs & abdomen — The combination of the ES of the lower limb muscles and the abdominal muscles.
  Arms: ES of limbs & abdomen

SUMMARY:
Background:

The presence of orthostatic hypotension (OH) as a consequence of blood volume redistribution during verticalisation in persons with spinal cord injury (SCI) is a common condition.

Aims:

To investigate the impact of three different types of electric stimulation (ES) (ES of the abdominal muscles versus ES of lower limb muscles versus simultaneously ES of abdominal and lower limb muscles versus control) on blood pressure stabilization and verticalisation-degrees between 0° and 70°. The hypothesis is, that the ES-induced contractions of the muscles cause a stabilisation respectively an increase of the blood pressure during the tilt-table test.

Subjects:

20 Women and men, at least 18 years of age, following an acute and traumatic SCI, with a lesion level above T6, an American Spinal Injury Association (AIS) Impairment Scale A,B or C and a diagnosis of OH (by tilt table test) were eligible for the study.

Methods:

Each patient underwent randomly three different types of ES sessions while being positioned on a tilt-table. The following sessions were planned:

A) ES of the abdominal muscles B) ES of the lower limb muscles C) Combination of A and B D) Control session (=diagnostic session)

Study type: Intervention Design: Prospective interventional study

ELIGIBILITY:
Inclusion Criteria:

* inpatients
* positive diagnosis of OH
* acute traumatic SCI
* lesion level above T6
* AIS A, B or C

Exclusion Criteria:

* fractures of the lower limbs
* decubitus (NPUAP >2)
* massive psychiatric dysfunction
* suicide intention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
blood pressure [mmHg] | 1 day (single measurement at each arm )

SECONDARY OUTCOMES:
Heart rate | 1 day (single measurement at each arm )

CONTACTS AND LOCATIONS:
Overall Officials: Aurelio Tobon, MD, Principal Investigator — Swiss paraplegic center
Locations (1):
- Swiss Paraplegic Center, Nottwil, Canton of Lucerne, Switzerland

REFERENCES:
- See also: Swiss Paraplegic Centre Nottwil — http://www.paraplegie.ch